CLINICAL TRIAL: NCT03570086
Title: Multiparametric Diagnostic Model of Thick-section Clinical-quality MRI Data in Detecting Migraine Without Aura
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xidian University (Other)
Responsible Party: Principal Investigator, Wei Qin, Professor, Xidian University
Other Study IDs: 20170908010418
Record Dates: First submitted 2018-05-28; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- migraineurs without aura
  Interventions: Diagnostic Test: diagnostic
- health controls
  Interventions: Diagnostic Test: diagnostic

INTERVENTIONS:
Diagnostic Test: diagnostic — using radiomics features from multiparametric thick-section clinical-quality brain MRI to distinguish migraineurs from health controls.

SUMMARY:
Recently, radiomics combined with machine learning method has been widely used in clinical practice. Compared with traditional imaging studies that explore the underlying mechanisms, the machine learning method focuses on classification and prediction to propose personalized diagnosis and treatment strategies. However, these studies were based on thin-section research-quality brain MR imaging with section thickness of < 2 mm. Clinical, the usage of thick-section clinical setting instead of thin-section research setting is especially important to shorten the acquisition time to reduce the patient's suffering. Here investigators want to build multiparametric diagnostic model of migraineurs without aura using radiomics features extracted from thick-section clinical-quality brain MR images.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* International Headache Society criteria for episodic migraine without aura

Exclusion Criteria:

* addition (including alcohol, nicotine, or drug)
* physical illness

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 200 migraineurs without aura 200 age- and gender-matched health controls (HCs)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
accuracy | 2018.7-2019.12
  a measure of statistical bias which measures the proportion of health controls and migrainures that are correctly identified as such.
sensitivity | 2018.7-2019.12
  true positive rate of detection in migraineurs which measures the proportion of actual migraineurs that are correctly identified as such.
specificity | 2018.7-2019.12
  true negative rate measures the proportion of actual health controls that are correctly identified as such.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China